CLINICAL TRIAL: NCT03025867
Title: Expanded Access Protocol for Niraparib in Patients With Recurrent Ovarian Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 3000-07-001
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

INTERVENTIONS:
Drug: Niraparib

SUMMARY:
This is an expanded access program (EAP) for eligible patients with Recurrent Ovarian Cancer.

This program is designed to provide access to niraparib prior to approval by the US Food and Drug Administration (FDA).

To be eligible, patients with Recurrent Ovarian Cancer following a partial (PR) or complete response (CR) to their most recent platinum-based chemotherapy and must have experienced a PR or CR after the penultimate (next to last) platinum-based chemotherapy for at least 6 months without disease progression after this chemotherapy.

DETAILED DESCRIPTION:
If a patient qualifies for participation in an ongoing niraparib clinical trial or is already participating in a niraparib clinical trial, she will not be able to participate in the EAP.

Ongoing clinical trials for niraparib include:

* A Phase 3 trial in patients who have received first-line treatment for ovarian cancer (the PRIMA trial, NCT # 02655016)
* A Phase 2 trial in patients who have received multiple lines of treatment for ovarian cancer (the QUADRA trial, NCT # 02354586)
* A Phase 1/2 trial in patients with advanced or metastatic triple-negative breast cancer or recurrent ovarian cancer. (the TOPACIO trial, NCT # 02657889)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
2. Completion of at least 2 previous courses of platinum-containing chemotherapy.
3. Had a CR or PR with duration of response >/=6 months following penultimate chemotherapy
4. Achieved a partial (PR) or complete (CR) tumor response following completion of the last platinum-containing chemotherapy [minimum of 4 cycles]
5. Patients previously treated with PARP inhibitors are eligible
6. Eastern Cooperative Oncology Group (ECOG, http://ecog-acrin.org/) performance status 0 or 1
7. Adequate organ function [Absolute neutrophil count (ANC) ≥ (greater than or equal to) 1,500/µL; Platelets ≥ (greater than or equal to) 100,000/µL; Hemoglobin ≥ (greater than or equal to) 9 g/dL]
8. Able to take oral medications
9. Women should not be pregnant at the beginning of the treatment and women or childbearing potential should not become pregnant while on niraparib
10. Patient should start treatment with niraparib no later than 12 weeks after completion of final dose of the platinum-containing chemotherapy

Exclusion Criteria:

1. Persistent ≥Grade 2 hematologic toxicity from prior cancer therapy
2. Known hypersensitivity to the components of niraparib
3. Patient is pregnant or breast feeding, or expecting to conceive children within the projected duration of the program treatment
4. Patient has uncontrolled hypertension

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult